CLINICAL TRIAL: NCT06852040
Title: Analysis of the Therapeutic Effect of TDCS Combined with Intraoral Electrical Stimulation on Dysphagia After Pontine Infarction
Brief Title: Effect of TDCS Combined with Intraoral Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuehai Lv (Other)
Responsible Party: Sponsor-Investigator, Xuehai Lv, Associate Chief Physician, Handan Central Hospital
Organization: Handan Central Hospital (Other)
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HandanCentral001
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pontine Infarction
Keywords: pontine infarction; dysphagia; transcranial direct current stimulation; Inductive electrical stimulation in the mouth
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group A (Active Comparator): A Swallowing neuromuscular electrical stimulator (LGT-2350A) from Guangzhou Longzhijie Medical Equipment Co., Ltd. was used. The electrodes are arranged sequentially on either side of the anterior midline of the neck. The parameter-selected electrical stimulation frequency is 80 Hz[12] (bidirectional square wave, pulse wave 300 microseconds, current intensity 10 to 25 mA） for 20 minutes each time, 1 time per day, 5 days/week, 4 weeks of treatment. which are limited to 20 min/time, 1 time/day, 5 days/week, and 4 weeks, respectively.
  Interventions: Device: Intraoral induction electrical stimulation therapy
- control group B (Active Comparator): tDCS treatment (specific method: microcurrent stimulator, stimulation electrode (3 cm×4 cm gelatin sponge), anodic stimulation site is the pharyngeal sensorimotor cortex area (between C3/T3 on the left[14], between C4/T4 on the right); the supraorbital area is the site of cathodic stimulation. The direct current intensity is 2.0 mA (20 min/time, 2 times/day) for two treatments (respectively, yin and yang alternating treatment), with an interval of at least 1 h, 5 days/week, and 4 weeks.
  Interventions: Device: tDCS treatment
- experimental group C (Experimental): tDCS combined with intraoral induction electrical stimulation. The patients were first treated with tDCS (the method is the same as that of the control group B) for 20 people twice a day and then given intraoral induction stimulation (the specific method is the same as that of the control group A) for 20 minutes, once a day, for 4 weeks.
  Interventions: Device: tDCS combined with intraoral induction electrical stimulation

INTERVENTIONS:
Device: Intraoral induction electrical stimulation therapy — Intraoral induction electrical stimulation therapy (specific method[13]: hand-held electrode rods were used to stimulate the mandibular hyoid muscle, digastric muscle, anterior abdomen, and other muscles of the three groups. Parameter setting: the frequency is 80Hz, the wave width is 1ms, the intensity is set to the muscle contraction, each electrical stimulation is 3s, intermittent 10s, 20min/time, 1 time/day, 5 days/week, 4 weeks is limited.
  Arms: control group A
Device: tDCS treatment — tDCS treatment (specific method: microcurrent stimulator, stimulation electrode (3 cm×4 cm gelatin sponge), anodic stimulation site is the pharyngeal sensorimotor cortex area (between C3/T3 on the left[14], between C4/T4 on the right); the supraorbital area is the site of cathodic stimulation. The direct current intensity is 2.0 mA (20 min/time, 2 times/day) for two treatments (respectively, yin and yang alternating treatment), with an interval of at least 1 h, 5 days/week, and 4 weeks.
  Arms: control group B
Device: tDCS combined with intraoral induction electrical stimulation — tDCS combined with intraoral induction electrical stimulation. The patients were first treated with tDCS (the method is the same as that of the control group B) for 20 people twice a day and then given intraoral induction stimulation (the specific method is the same as that of the control group A) for 20 minutes, once a day, for 4 weeks.
  Arms: experimental group C

SUMMARY:
Objective: To investigate the clinical efficacy of transcranial direct current stimulation (tDCS) combined with intraoral electrical stimulation in patients with dysphagia after pontine infarction. Methods: This prospective study enrolled a total of 90 patients with dysphagia due to pontine infarction from October 2022 to November 2024, and they were divided into three groups according to the treatment method: control group A, control group B, and experimental group C. Control group A was given intraoral induction electrical stimulation, control group B was given transcranial direct current stimulation (tDCS), and experimental group C was given tDCS combined with intraoral induction electrical stimulation. The three groups were compared in terms of efficacy, modified Waffield Drinking Water Test Score (MWST), Penetration-aspiration scale (PAS), Functional Oral Intake Scale (FOIS), Hyoid-Larynx Complex mobility, maximum amplitude of surface electromyography, and swallowing time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysphagia (able to cooperate with swallowing assessment) and consistent with the criteria of the "Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018"[9] or pontine infarction by clinical imaging examination;
* Age≥18 years or ≤80 years;
* The modified water swallow test (MWST) score is 3-5[10] or the Functional Oral Intake Scale score <4

Exclusion Criteria:

* Those who are intolerant to electrical stimulation or allergic to auxiliary electrodes;
* Patients with implanted pacemakers, metal stents in the neck, or other reasons that cannot be treated with electrical stimulation;
* Patients who are critically ill or unable to cooperate with the assessment and treatment of patients with dysphagia due to other reasons.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
MWST | 4 weeks
  The patient was instructed to stay in a Sitting or standing position, drink 1 ml, 3 ml, and 5 ml of water, respectively, and drink 30 ml of water when the patient did not show abnormal manifestations. The severity of dysphagia is classified as 1-5 according to the time the patient drinks water, whether there is choking, swallowing in fractions, etc., and the lower the rating, the better the swallowing function. (1) significantly effective: the MWST assessment reached grade 1 or decreased ≥ grade 2. (2) Effective: MWST assessment is reduced by 1 level. (3) Ineffective: There is no change before and after the MWST assessment. Total effective rate = (significant effect + effective) number of cases/total number x 100%.
FOIS | 4 weeks
  The patient's oral feeding function is according to the type of food and the way the patient eats. 1 point: No oral food at all; 2 points: Dependent on tube feeding, can try to eat the smallest amount; 3 points: 3 points: tube feeding, oral ingestion of food or liquid of single quality；4 points: Completely oral consumption of a single quality of food; 5 points: Completely oral consumption of a variety of food qualities, but special preparation or compensation is required; 6 points: Eat completely by mouth, but with special food restrictions; 7 points: No restriction on complete oral feeding, The score is directly proportional to the swallowing function.
RAS | 4 weeks
  1 point, the bolus does not enter the airway; 2 points, the bolus enters the airway, is above the level of the vocal cords, and is ejected from the airway; 3 points, the bolus enters the airway, is above the level of the vocal cords, and is not ejected from the airway; At 4 minutes, the bolus enters the airway and is ejected from the airway; 5 points, the bolus enters the airway, but does not eject from the airway; 6 points, the substance enters the airway, reaches below the level of the vocal cords, and is ejected into the larynx or outside the airway; At 7 minutes, the bolus enters the airway and reaches below the level of the vocal cords, but the force is still not ejected from the trachea; At 8 points, the bolus enters the airway, reaches below the level of the vocal cords, and is unable to eject. PAS was assessed according to the Videofluoroscopy Swallowing Study (VFSS) or Point-of-Care Fiberoptic Endoscopic Swallowing.
Hyoid laryngeal complex mobility | 4 weeks
  X-ray recording of the upward and anterior displacement of the hyoid bone and thyroid cartilage during swallowing. After 4 weeks of treatment, the dynamic (swallowing state), the static hyoid bone, and thyroid cartilage positions, and the dynamic and static differences of thyroid cartilage and hyoid bone in the vertical and horizontal directions were recorded as the upward distance and forward distance, respectively.
Maximum Amplitude and Swallowing Time of Surface Electromyography | 4 weeks
  Maximum Amplitude: This refers to the highest voltage peak recorded by the electromyography (EMG) analyzer during the swallowing process. It is an indicator of the strength of muscle activation involved in swallowing. Higher maximum amplitudes suggest stronger muscle contractions and potentially better swallowing function.Swallowing Time: This is the duration, measured in seconds, from the onset of the swallowing action (initiated by the movement of the tongue) to the completion of the bolus passing through the pharynx and entering the esophagus. Shorter swallowing times are generally associated with more efficient swallowing mechanics and reduced risk of aspiration.

CONTACTS AND LOCATIONS:
Overall Officials: Xuehai Lv Lv, Principal Investigator — Handan Central Hospital
Locations (1):
- Handan Central Hospital, Handan, Hebei, China

IPD SHARING:
Plan to Share IPD: No